CLINICAL TRIAL: NCT06894719
Title: Prolonged Oral Tranexamic Acid Use in Primary Total Joint Arthroplasty: A Double Blind Randomized Placebo Controlled Trial
Brief Title: Oral Tranexamic Acid After Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Bailey Terhune, Principle Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25031706
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Arthroplasty
Keywords: tranexamic acid; range of motion; postoperative pain; postoperative function
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized via computer-generated assignment and remain blinded to treatment. Data collection includes ROM assessments at follow-ups, surveys, and chart reviews for complications. This study aims to optimize oral TXA dosing in TKA to improve recovery while maintaining safety and cost-effectiveness.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral-Short Arm: 1.95g TXA daily POD 1-3 (Active Comparator): 1.95g TXA daily for post operative days 1-3
  Interventions: Drug: tranexamic acid Oral-Short Arm
- Oral-Long Arm (Active Comparator): 1.95g TXA daily for post operative days 1-7
  Interventions: Drug: tranexamic acid Oral-Long Arm
- Control Group: Placebo for 3 days post-op (Placebo Comparator): Placebo for 3 days post-op
  Interventions: Drug: Control group placebo

INTERVENTIONS:
Drug: tranexamic acid Oral-Short Arm — 1.95g Tranexamic acid daily for post op days 1 to 3
  Arms: Oral-Short Arm: 1.95g TXA daily POD 1-3
Drug: tranexamic acid Oral-Long Arm — 1.95g tranexamic acid daily post op days 1-7
  Arms: Oral-Long Arm
Drug: Control group placebo — Placebo for 3 days post-op
  Arms: Control Group: Placebo for 3 days post-op

SUMMARY:
This is a prospective, double-blind, randomized controlled trial evaluating the efficacy of oral tranexamic acid (TXA) in total knee arthroplasty (TKA). The study will assess pain, function, and range of motion (ROM) over a 2-year period, with key evaluations at 6 weeks and 90 days postoperatively.

Hypothesis:

Patients receiving 1.95g oral TXA for 3 or 7 days post-op will show improved pain, function, and ROM at 6 weeks and 90 days, with similar blood loss and transfusion rates as the control group.

DETAILED DESCRIPTION:
OBJECTIVES:

Purpose:

This is a prospective, double-blinded, randomized control study to evaluate the efficacy and role of oral Tranexamic acid in total knee arthroplasty by assessing pain, function, and range of motion over a 2-year follow-up period.

Hypothesis:

We hypothesize that those given 1.95g oral TXA for 3- and 7-days post-op will have improved pain, function, and range of motion assessed at the 6-week follow-up along with improved range of motion (ROM) at the 90-day follow-up. Additionally, we expect both the control group and the experimental group to have similar blood loss and transfusion rates.

BACKGROUND:

As the rates of primary and revision total knee arthroplasty (TKA) continue to rise in the United States2,3, it is more important than ever to evaluate and improve primary and secondary outcomes as well as costs associated with these procedures. Tranexamic acid (TXA) has been widely used to improve morbidity and mortality in TKA, with substantial evidence demonstrating its efficacy in reducing blood loss6,7,11,12,13 and transfusion rates6,7,12. A meta-analysis done by Drain et al. also showed a significant reduction in periprosthetic joint infection (PJI) and length of stay4,12 in patients receiving any form of intraoperative TXA. Subsequent studies confirmed that TXA is safe for use in TKA, as it does not increase the incidence of complications including thromboembolic events and renal failure, even in high-risk populations5,6.

Recent literature has increasingly focused on comparing oral versus intravenous (IV) TXA in TKA, aiming to reduce costs while maintaining comparable safety and efficacy to the intravenous formulation. Current evidence strongly supports the noninferiority of preoperative oral TXA compared to IV TXA 8,9,10,14. Similar findings have been reported in revision TKA1. However, a key limitation of these studies is that their primary outcomes are often confined to blood loss, transfusion rates, thromboembolic events, and length of stay. Additionally, significant variability exists in the dosage regimens used across these studies.

While previous research has explored different formulations, doses, and delivery timings of TXA1,7,15, there is limited data on the optimal dosing strategy and length of administration for oral TXA. Most studies focus on perioperative administration, with few investigating the use of TXA beyond postoperative day one16,18,19. Some evidence supports extended IV TXA use for improving clinical parameters such as hemoglobin levels, though further research is needed18,19,20.

Currently, there is a lack of literature examining extended oral TXA use in primary TKA. Existing studies have produced conflicting results regarding pain and function outcomes16,21, with inconsistent dosing regimens further complicating efforts to draw firm conclusions.

Further evaluation of oral TXA administration during the perioperative period and beyond could provide valuable insights for enhancing the safety and reducing the costs of outpatient TKA. Establishing an optimal standard oral dose for prolonged TXA use could improve outcomes, support the transition to outpatient care, and provide consistent post-discharge management protocols.

The purpose of this study is to evaluate the efficacy and role of oral TXA in primary TKA by assessing pain, function, and range of motion over a 2-year follow-up period. We hypothesize that mid-term improvements in pain, function, and range of motion will be observed, with improved clinical outcomes such as arch of motion at the 2-year mark.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary TKA at Rush main hospital or participating ASC
* Willingness to undergo randomization to take medication potentially up to 7 days post op.
* Willing to answer daily questions on pain, functionality and opioid consumption

Exclusion Criteria:

* History of venous thromboembolism, MI, or stroke in the past year
* Patients on any chronic anticoagulation medications besides Aspirin
* Patients with Cancer
* Patients with end stage renal disease that are on dialysis
* Drug allergy to TXA
* Taking oral birth control
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: knee range of motion | (flexion/extension) at 2 weeks and 6 weeks post op
  Primary Endpoint:
  Knee ROM

SECONDARY OUTCOMES:
Secondary" VAS pain scores | 2 weeks, 6 weeks, and 3 months post op
  Pain scores (VAS)
Secondary: KOOS Jr | 2 weeks. 6 weeks, 3 months post op
secondary: EQ-5D-3L functional scores | 2 weeks, 6 weeks, and 3 months post op
Adverse events and complications | 3 months post op
  Any adverse events or complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bailey Terhune, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, once all participants have completed all parts of the study
Supporting Information: Study Protocol, SAP
Time Frame: 6 months following end of study and will last for a year
Access Criteria: unending